CLINICAL TRIAL: NCT03456037
Title: Incidence Of Hepatitis And Its Effect On Prognosis In Patients Who Follow In Intensive Care Unit
Brief Title: Incidence Of Hepatitis In Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, Assistant Professor, Sakarya University
Other Study IDs: hepatitis
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Intensive Care Unit
Keywords: HBsAg; Anti-HCV,; seropositivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: hepatitis viruses — There are 5 main hepatitis viruses, referred to as types A, B, C, D and E. These 5 types are of greatest concern because of the burden of illness and death they cause and the potential for outbreaks and epidemic spread. In particular, types B and C lead to chronic disease in hundreds of millions of people and, together, are the most common cause of liver cirrhosis and cancer.The aim is to investigate incidence of HBsAg, anti-HCV in serum samples and evaluation of biomarkers taken from patients who were followed the intensive care unit of Sakarya University Training and Research Hospital.

SUMMARY:
The aim is to investigate incidence of HBsAg, anti-HCV in serum samples and evaluation of biomarkers taken from patients who were followed the intensive care unit of Sakarya University Training and Research Hospital and The intensive care unit attracts attention by making health workers more susceptible to the risk of hepatitis.

DETAILED DESCRIPTION:
This retrospective study included 536 cases who were followed with various diagnoses in intensive care units between 1 Ocak 2015 ile 1 Ocak 2016, covering the six months period, retrospectively. Sakarya University's Faculty of Medicine Review Board (71522473/050.01.04/113) approved the study after approval of the research ethics committee (. Medical record forms and electronic medical record system of the hospital were used in the analysis of medical data with regard to age, sex, HBsAg, anti-HCV, AST, ALT, bilirubin, creatinine levels.

ELIGIBILITY:
Inclusion Criteria:

All patients who were followed in the intensive care unit

Exclusion Criteria:

None

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted from 1 january 2015 to 1 january 2016 . Patients who were followed with various diagnoses in intensive care units between 1 january 2015 to 1 january 2016, covering the one year period, retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
HBsAg | 1 month
  HBsAg is the serologic hallmark of HBV infection and is the first marker to appear after acute infection.

SECONDARY OUTCOMES:
anti-HCV | 1mounth
  Anti-HCV antibody tests look for antibodies to HCV in the blood, indicating an HCV infection has occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Sayhan,, Assis Prof, Study Chair — Sakarya University Research and Training Hospital
Locations (1):
- Sakarya University Research and Training Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dayan S, Tekin A, Tekin R, Dal T, Hosoglu S, Yazgan UC, Bekcibasi M, Gul K. HBsAg, anti-HCV, anti-HIV 1/2 and syphilis seroprevalence in healthy volunteer blood donors in southeastern Anatolia. J Infect Dev Ctries. 2013 Sep 16;7(9):665-9. doi: 10.3855/jidc.2835. PMID 24042102